CLINICAL TRIAL: NCT07243093
Title: Validating a Deep Learning Algorithm in Children With Ear Concerns
Brief Title: Validating and AI Software for Assessment of Children With Ear Concerns
Status: Not yet recruiting | Type: Observational
Sponsor: Glimpse Diagnostics, Inc. (Industry)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); Clinical Research Strategies (Unknown)
Responsible Party: Sponsor
Other Study IDs: Glimpse-01; 1R44EB036883-01A1 (NIH)
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Otalgia; Otitis Media; Otitis Media Effusion
MeSH Terms: conditions — Earache; Otitis Media; Otitis Media with Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

SUMMARY:
The goal of this observational study is to determine if the Glimpse machine learning algorithm can accurately assess ear diseases in children. Participants will:

* Have a video of their ear taken by their parent or their guardian
* Have a video of their ear taken by a Primary Care Physician (PCP)
* Have an assessment of their eardrums and a video of their ears taken by an Ear, Nose, and Throat specialist (ENT).

The videos will be used to determine if the Glimpse algorithm matches the diagnosis of the physicians.

DETAILED DESCRIPTION:
Ear complaints, including earache (otalgia), are the most common reasons children seek healthcare and routinely bring children into the office of a pediatrician or urgent care setting. This study will assess children who present with signs and symptoms of otitis media to the primary care office or urgent care. Participants will receive their standard of care from their treating physician, with study assessments including videos of their ears taken by their parent or guardian and the treating physician. Once this is complete, participants will see an ENT for an assessment of their eardrum. The ENT assessment will occur within 24 hours of the PCP visit and will not be used to inform patient treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 6 months to 6 years
* Presenting to a pediatrician's office or urgent care with signs and symptoms of otitis media, including tugging at ears, ear pain, crying at night, refusing to lie flat, sleeping poorly, having a fever, having decreased appetite, and/or concern for hearing loss, regardless of previous diagnosis of AOM or OME.

Exclusion Criteria:

* History of craniofacial abnormality
* PE tubes currently in place
* Current otorrhea
* Caretaker not having use of both hands and arms

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 6 months to 6 years presenting with ear concerns
Sampling Method: Non-Probability Sample
Enrollment: 658 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Percent agreement of Glimpse machine learning algorithm's classification of a child's ear image with an ENT panel diagnosis | Within 24 hrs of presenting to PCP or urgent care office
  The primary endpoint of this study is to compare the percent agreement of Glimpse machine learning algorithm's classification of a child's ear image with an ENT panel diagnosis of the same child's ear for the diagnoses of acute otitis media (AOM), otitis media with effusion (OME), and no middle ear effusion, versus the percent agreement of primary care provider's (PCP) diagnosis with an ENT panel diagnosis, of in children with otalgia.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bryton C, Surapaneni S, Rangarajan N, Hong A, Marston AP, Vecchiotti MA, Hill C, Scott AR. Deep learning algorithm classification of tympanostomy tube images from a heterogenous pediatric population. Int J Pediatr Otorhinolaryngol. 2025 May;192:112311. doi: 10.1016/j.ijporl.2025.112311. Epub 2025 Mar 13. PMID 40096786